CLINICAL TRIAL: NCT06139081
Title: The Effect of Different Oxygen Delivery Methods of Nasal Catheter on the Incidence of Hypoxemia in Patients with High Risk of Hypoxia During Painless Gastroscopy
Brief Title: Oxygen Delivery Methods of Nasal Catheter on the Incidence of Hypoxemia in Patients with Painless Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20230915-10
Record Dates: First submitted 2023-10-26; First posted 2023-11-18 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Transnasal oxygen was administered by nasal catheter before gastroscopy, transoral oxygen was administered by nasal catheter during gastroscopy, and transnasal oxygen was administered by nasal catheter after withdrawal of gastroscope.
  Interventions: Other: Oxygen delivery mode
- Group B (No Intervention): Nasal catheter was used to give oxygen before, during and after withdrawal of gastroscope

INTERVENTIONS:
Other: Oxygen delivery mode — After the implantation of the mirror, nasal catheter was used to give oxygen through the mouth
  Arms: Group A

SUMMARY:
In this study, patients undergoing painless gastroscopy were selected to change the nasal catheter oxygen delivery mode to oral oxygen delivery after endoscope implantation, in order to explore the effect of this oxygen delivery mode on the incidence of hypoxemia during general anesthesia gastroscopy.

DETAILED DESCRIPTION:
This study was a randomized controlled study in which patients undergoing elective painless gastroscopy were selected and grouped by random number table. The control group used conventional nasal cannula oxygen method: nasal cannula was used before, during and after gastroscopy was implanted and after withdrawing from the gastroscopy. Test group: Before the gastroscope enters the oral cavity, oxygen is administered through a nasal catheter via the nose. After the gastroscope enters the oral cavity, oxygen is administered through the nasal catheter via the mouth. After the gastroscope is withdrawn, oxygen is administered through the nasal catheter via the nose. The incidence of intraoperative hypoxemia was observed.

ELIGIBILITY:
Inclusion Criteria:

Patients who receiving gastroscopy under general anesthesia, accompanied with one of the following risk factors of hypoxia:

1. Patients combined with heart or respiratory diseases
2. Age older than 60
3. ASA grading II-III
4. BMI≥30kg/m²,
5. Snoring or having sleep apnea syndrome
6. Patients with a STOP-Bang score ≥ 3 (the risk of OSAS is high) are considered to be highly risk of hypoxia.

Exclusion Criteria:

1. Severe cardiovascular, pulmonary, liver, or kidney disease
2. Patients with infections or tumors of airway
3. History of difficult intubation under general anesthesia
4. Severe sleep apnea syndrome [hypopnea/apnea hypopnea index (AHI)>40]
5. Patients allergic to propofol, eggs, soy or egg whites
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxemia | Five minutes after finishing gastroscopy examination
  SpO2<92%

CONTACTS AND LOCATIONS:
Overall Officials: Gu Jianping, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tas Z, Hosten T, Kus A, Cesur S, Turkyilmaz N, Arikan A, Solak ZM. Comparison of tidal volume and deep breath preoxygenation techniquesundergoing coronary artery bypass graft surgery: effects of hemodynamicresponse and arterial oxygenation. Turk J Med Sci. 2017 Nov 13;47(5):1576-1582. doi: 10.3906/sag-1606-132. PMID 29151335
- [Background] Chen DX, Yang H, Wu XP, Niu W, Ding L, Zeng HL, Li Q. Comparison of a Nasal Mask and Traditional Nasal Cannula During Intravenous Anesthesia for Gastroscopy Procedures: A Randomized Controlled Trial. Anesth Analg. 2022 Mar 1;134(3):615-623. doi: 10.1213/ANE.0000000000005828. PMID 34878412
- [Background] Gavrilovska-Brzanov A, Shosholcheva M, Kartalov A, Jovanovski-Srceva M, Brzanov N, Kuzamanovska B. Medium-Flow Oxygenation Through Facial Mask and Nasal Cannula in a Limited Resource Setting. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2022 Jul 13;43(2):101-109. doi: 10.2478/prilozi-2022-0023. PMID 35843919